Comparison between inhalational anesthetic (sevoflurane) and intravenous anesthetic (propofol infusion) for maintenance of sedation during Endoscopic retrograde cholangiopancreatography

Principle investigator
Dr. Vijai Kumar
Senior Lecturer

Department of Anesthesiology SIUT Karachi

Dated: 01-07-2021

## **DATA ANALYSIS:**

For data analysis SPSS software will be used of version 22. Mean and standard deviation will be computed for variable such as age, height, BMI, RSS, HR, SBP, DBP and MAP at 0,1,3,5,10 min. For determining the differences in the hemodynamics mean unpaired "t" test will be used between groups. Categorically Variables such as gender, ASA and post op complications like gagging, PONV, Apnea and cough will be presented as frequencies and percentages.

Chi-square test will be followed and used between 2 groups, there proportion difference will be compared using P value

(Note: This plan is a part of synopsis which we have uploaded on NCT form)



SIUT SINDH INSTITUTE OF UROLOGY AND TRANSPLANTATION

Approval No: SIUT-ERC-2021/A-325

Approval Issued: August 30, 2021

Vijay Kumar Department of Anesthesia, SIUT

Re: <u>Project Title "Comparison between inhalational anesthetic (sevoflurane) and intravenous anesthetic (propofol infusion) for maintenance of sedation during Endoscopic retrograde cholangiopancreatography."</u>

Dear Dr. Vijay Kumar,

Thank you for submitting the above referenced protocol to the SIUT-Ethical Review Committee (ERC). ERC finds that this protocol raises no ethical concerns. Approval is granted and you may commence your research. According to SIUT-ERC requirements, the ERC approval number should be clearly printed and visible on all consent forms used in the study.

Please note that this approval is valid for one year and relates to the ethical content of the study only. If you make any changes to the protocol during the period of this approval, you must submit a revised protocol to the SIUT-ERC for approval before implementing the changes.

SIUT-ERC requires a follow up from all researchers about the status of the approved research at the completion of one year from the date of issuance. You are also expected to comply with this practice.

Yours Sincerely,

Ali Lanewala, DABIM, DABP, DAB Nephrology Professor and In charge Pediatric Nephrology, Co-Chair, SIUT-Ethical Review Committee (SIUT-ERC)